CLINICAL TRIAL: NCT02317744
Title: Treatment of Binge Eating Disorder in Obesity: Naltrexone/ Bupropion Combination Versus Placebo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1409014705
Record Dates: First submitted 2014-12-11; First posted 2014-12-16 (Estimated); Results first posted 2017-12-22 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-11

CONDITIONS: Binge Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder | interventions — Naltrexone-Bupropion combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Naltrexone/ Bupropion combination (Experimental): 50 mg naltrexone and 300 mg bupropion per day for 3 months
  Interventions: Drug: Naltrexone and bupropion combination
- Pill placebo (Placebo Comparator): Daily placebo medication for 3 months
  Interventions: Other: Pill Placebo

INTERVENTIONS:
Drug: Naltrexone and bupropion combination
  Arms: Naltrexone/ Bupropion combination
Other: Pill Placebo
  Arms: Pill placebo

SUMMARY:
This study will test the effectiveness of the combination of Naltrexone and Bupropion relative to placebo for reducing binge eating in persons with obesity and binge eating disorder.

ELIGIBILITY:
Inclusion Criteria:

* Binge eating disorder (full criteria as described in the American Psychiatric Association Diagnostic and Statistical Manual of Mental Disorders, 5th edition)
* BMI between 30 kg/m2 and 50 kg/m2
* Not taking anti-depressant medications
* Read English proficiently enough to read study assessments
* Available for duration of treatment plus follow-up period
* Able to travel to study location (New Haven, CT) for monthly visits
* Agree to study procedures

Exclusion Criteria:

* Medical status judged by study physician as contraindication
* History of seizures
* Past or current anorexia nervosa, bulimia nervosa
* Current medications that influence eating/weight
* Current substance use disorder or other severe psychiatric disturbance (e.g., suicidality) that requires immediate treatment
* Pregnant or breastfeeding

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos M Grilo, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Grilo CM, Lydecker JA, Morgan PT, Gueorguieva R. Naltrexone + Bupropion Combination for the Treatment of Binge-eating Disorder with Obesity: A Randomized, Controlled Pilot Study. Clin Ther. 2021 Jan;43(1):112-122.e1. doi: 10.1016/j.clinthera.2020.10.010. Epub 2020 Nov 18. PMID 33218742

RESULTS

PARTICIPANT FLOW:
Groups:
- Naltrexone/ Bupropion Combination: 50 mg naltrexone and 300 mg bupropion per day for 3 months
  Naltrexone and bupropion combination
- Pill Placebo: Daily placebo medication for 3 months
  Pill Placebo
Period: Overall Study
Arm/Group | Naltrexone/ Bupropion Combination | Pill Placebo
Started | 12 | 10
Completed Treatment | 10 | 7
Completed | 11 (One NB participant stopped the treatment but completed assessments.) | 8 (One Placebo participant stopped the treatment but completed assessments.)
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone/ Bupropion Combination | Pill Placebo | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 10 | 22
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (8.0) | 49.4 (10.1) | 50.4 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 10 | 22
Binge Eating Frequency [Mean (Full Range); unit: binge eating days (out of 28)] | 16.0 [4 to 28] | 9.2 [3 to 27] | 12.9 [3 to 27]
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] | 35.0 [30 to 49] | 40.1 [33 to 48] | 37.3 [30 to 49]

OUTCOME MEASURES:

1. Primary Outcome: Binge Eating Frequency (Continuous)
Description: Binge eating will be assessed by interview and self-report and the primary outcome is frequency. Frequency also is defined continuously (analyzed dimensionally).
Time Frame: Post-treatment (at 3 months)
Measure: Mean (Full Range); unit: binge eating days (out of 28)
Arm/Group | Naltrexone/ Bupropion Combination | Pill Placebo
Number analyzed (Participants) | 11 | 8
binge eating days (out of 28) | 4.4 [0 to 28] | 3.0 [0 to 16]

2. Primary Outcome: Binge Eating Frequency (Continuous)
Description: as for outcome 1
Time Frame: 6 month follow-up (an average of 6 months following treatment)
Measure: Mean (Full Range); unit: binge eating days (out of 28)
Arm/Group | Naltrexone/ Bupropion Combination | Pill Placebo
Number analyzed (Participants) | 8 | 8
binge eating days (out of 28) | 5.4 [0 to 25] | 2.9 [0 to 14]

3. Secondary Outcome: Body Mass Index (BMI)
Description: BMI is calculated using measured height and weight.
Time Frame: Post-treatment (at 3 months)
Measure: Mean (Full Range); unit: kg/m^2
Arm/Group | Naltrexone/ Bupropion Combination | Pill Placebo
Number analyzed (Participants) | 11 | 9
kg/m^2 | 34.5 [29 to 48] | 39.7 [32 to 47]

4. Secondary Outcome: Body Mass Index (BMI)
Description: BMI is calculated using measured height and weight.
Time Frame: 6 month follow-up (an average of 6 months following treatment)
Measure: Mean (Full Range); unit: kg/m^2
Arm/Group | Naltrexone/ Bupropion Combination | Pill Placebo
Number analyzed (Participants) | 8 | 8
kg/m^2 | 35.9 [28 to 48] | 40.3 [34 to 45]

ADVERSE EVENTS:
Time Frame: 3 months
Description: Participants were interviewed by research clinicians monthly during treatment (3 months) about the absence or presence of side effects.
Arm/Group | Naltrexone/ Bupropion Combination | Pill Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/8
Other Adverse Events (participants affected / at risk) | 11/11 | 5/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Naltrexone/ Bupropion Combination (N=11) | Pill Placebo (N=8)
Anxiety (Psychiatric disorders) | 3 | 5 — 1 participant discontinued NB because of anxiety; 1 participant discontinued placebo because of anxiety.
Vomiting (Gastrointestinal disorders) | 3 | 0 — 1 participant discontinued NB because of vomiting; 0 participants discontinued placebo because of vomiting.
Constipation (Gastrointestinal disorders) | 2 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 2
Dizziness (General disorders) | 5 | 1
Dry Mouth (General disorders) | 2 | 2
Headache (General disorders) | 3 | 4
Insomnia (General disorders) | 5 | 1
Nausea (Gastrointestinal disorders) | 5 | 2
Hot Flush (General disorders) | 4 | 1
Fatigue (General disorders) | 2 | 1
Common Cold (General disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 1
Sinusitis (General disorders) | 0 | 1
Sexual Dysfunction (General disorders) | 0 | 0
Depression (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No